CLINICAL TRIAL: NCT03520322
Title: A Prospective, Randomized, Blinded, Placebo-controlled, Single Center, Efficacy Study of a Mastoid Device in Subjects With Ménière's Disease
Brief Title: A Study of a Mastoid Device in Subjects With Ménière's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RSRB 63989
Record Dates: First submitted 2018-04-27; First posted 2018-05-09 (Actual); Results first posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Meniere Disease
MeSH Terms: conditions — Meniere Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Mastoid Oscillator (Experimental): patients with Menieres Disease
  Interventions: Device: Mastoid Oscillator
- Control device (Placebo Comparator): patients with Menieres Disease
  Interventions: Device: Control Device

INTERVENTIONS:
Device: Mastoid Oscillator — The oscillator will be placed over the mastoid of their involved ear and secured via an elastic/Velcro headband. The subject is positioned so as to place the endolymphatic duct into a gravitationally dependent orientation (the subject lying on their contralateral side with the face slightly tilted towards the floor). The device is turned on and operated for 30 minutes.
  Arms: Mastoid Oscillator
Device: Control Device — The control device will be placed over the mastoid of their involved ear and secured via an elastic/Velcro headband. The subject is positioned so as to place the endolymphatic duct into a gravitationally dependent orientation (the subject lying on their contralateral side with the face slightly tilted towards the floor). The device is turned on and operated for 30 minutes.
  Arms: Control device

SUMMARY:
The purpose of this study is to investigate the efficacy of a mastoid treatment device in patients with active Ménière's disease that is not controlled by traditional medical management

DETAILED DESCRIPTION:
This is a single center, randomized, placebo-controlled trial of mastoid oscillation for treatment of Ménière's disease. Eligible subjects will be randomized using a 1:1 allocation to either mastoid oscillation or placebo (oscillator device that provides the same sound but no vibration of the mastoid) received for 30 minutes at four weekly study visits, with efficacy determination via change in frequency and severity of Ménière's symptoms following the final study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 and older
2. Clinical diagnosis of Ménière's disease, with classical symptoms:

i. Episodic spinning vertigo ii. Fluctuating unilateral low frequency sensorineural hearing loss iii. Tinnitus iv. Aural fullness c. Failure of traditional medical management of Ménière's disease symptoms d. English language skills sufficient to provide informed consent to the study

Exclusion Criteria:

1. Atypical medical history of Ménière's symptoms and questionable Ménière's diagnosis
2. Bilateral Ménière's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-12-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- 2365 S. Clinton Ave, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject was consented but not randomized to the intervention.
Period: Overall Study
Arm/Group | Mastoid Oscillator | Control Device
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mastoid Oscillator | Control Device | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in the Number of Monthly Vertigo Episodes
Description: A patient reported measure of the number of vertigo episodes they have experienced in the past month.
Time Frame: Baseline to 90 days
Measure: Mean (Standard Deviation); unit: Episodes per month
Arm/Group | Mastoid Oscillator | Control Device
Number analyzed (Participants) | 3 | 3
Episodes per month | 20.8 (26) | 22.2 (4.8)

2. Secondary Outcome: Change in Average Pure Tone Threshold
Description: The audiometric thresholds measured at 500 Hz, 1, 2, & 4 kHz under controlled conditions are averaged together to create the average pure tone threshold
Time Frame: Baseline to 90 days
Measure: Mean (Standard Deviation); unit: Decibels
Arm/Group | Mastoid Oscillator | Control Device
Number analyzed (Participants) | 3 | 3
Decibels | 6.0 (16.6) | 5.4 (7.8)

3. Secondary Outcome: Change in Percentage of Words Recognized
Description: A standard audiological evaluation of the percentage of words recognized from a list of 50 when played under controlled conditions
Time Frame: Baseline to 90 days
Measure: Mean (Standard Deviation); unit: percentage of words
Arm/Group | Mastoid Oscillator | Control Device
Number analyzed (Participants) | 3 | 3
percentage of words | -8.7 (12) | 1.3 (6.5)

4. Secondary Outcome: Change in Meniere's Functional Level
Description: A patient reported measure of their overall function from 0 to 6 where 0 corresponds to no symptoms and 6 corresponds to completely debilitated.
Time Frame: Baseline to 90 days
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mastoid Oscillator | Control Device
Number analyzed (Participants) | 3 | 3
Score on a scale | -1 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: 90 days
Description: Adverse events defined as discomfort related to the treatment were collected. In addition, subject electronic health records were reviewed for mortality or potential AEs at the end of the study.
Arm/Group | Mastoid Oscillator | Control Device
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-07): https://cdn.clinicaltrials.gov/large-docs/22/NCT03520322/Prot_SAP_000.pdf